CLINICAL TRIAL: NCT00616239
Title: The Efficacy of Salicylic Acid Peels Combined With 4% Hydroquinone Cream Versus 4% Hydroquinone Cream Alone in the Treatment of Hispanic Women With Moderate to Severe Melasma
Brief Title: Salicylic Acid Peels Combined With 4% Hydroquinone in the Treatment of Moderate to Severe Melasma in Hispanic Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Amit Pandya, Professor of Dermatology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 082007-078; IRB File 082007-078
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Melasma
Keywords: Melasma; Dark spots on the face
MeSH Terms: conditions — Melanosis | interventions — Chemexfoliation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Subjects randomized to have the right side of the face peeled with salicylic acid every 2 weeks for a total of 4 peels (first 2 at 20% and last 2 at 30%). Subjects will apply 4% hydroquinone cream to affected areas on entire face for 14 weeks.
  Interventions: Drug: 20-30% Salicylic Acid peels to the right side of the face
- B (Active Comparator): Subjects randomized to have the left side of the face peeled with salicylic acid every 2 weeks for a total of 4 peels (first 2 at 20% and last 2 at 30%). Subjects will apply 4% hydroquinone cream to affected areas on entire face for 14 weeks.
  Interventions: Drug: 20-30% Salicylic Acid peels to the left side of the face

INTERVENTIONS:
Drug: 20-30% Salicylic Acid peels to the right side of the face — Two 20% salicylic acid peels two weeks apart followed by 2 30% salicylic acid peels two weeks apart to the right side of the face.
  Other Names: Chemical Peels
  Arms: A
Drug: 20-30% Salicylic Acid peels to the left side of the face — Two 20% salicylic acid peels two weeks apart followed by 2 30% salicylic acid peels two weeks apart to the left side of the face
  Other Names: Chemical Peels
  Arms: B

SUMMARY:
This study will enroll 20 adult Hispanic women. Participants will apply 4% hydroquinone cream twice daily to affected areas on the face for 14 weeks and half the face will be peeled with 20-30% salicylic acid every two weeks for a total of 4 peels. The first two peels will be 20% salicylic acid and the second two peels will be with 30% salicylic acid. The purpose of the study will be to evaluate the safety and efficacy of salicylic acid combined with 4% hydroquinone versus 4% hydroquinone alone.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic women ages 18-65 years of age with moderate to severe melasma
* English and Spanish-speaking women

Exclusion Criteria:

* Pregnant or breast-feeding women
* Subjects who have used 4% hydroquinone within 3 months of study start
* Subjects who have used chemical peels, microdermabrasion or facial laser treatments within 9 months of study start

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Pandya, M.D., Principal Investigator — UT Southwestern Medical Center at Dallas - Department of Dermatology
Locations (1):
- UT Southwestern Medical Center at Dallas - Dermatology Clinical Trials, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 20% to 30% Salicylic Acid Peels + 4% Hydroquinone Cream: Subjects randomized to have the right side of the face peeled with salicylic acid every 2 weeks for a total of 4 peels (first 2 at 20% and last 2 at 30%). Subjects will apply 4% hydroquinone cream to affected areas on entire face for 14 weeks.
Period: Overall Study
Arm/Group | 20% to 30% Salicylic Acid Peels + 4% Hydroquinone Cream
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | 20% to 30% Salicylic Acid Peels + 4% Hydroquinone Cream
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing Improvement of Melasma Based on Mexameter Readings
Description: Improvement of melasma on the peel side using mexameter reading
Time Frame: 14 weeks
Measure: Number; unit: participants
Arm/Group | 20% to 30% Salicylic Acid Peels + 4% Hydroquinone Cream
Number analyzed (Participants) | 18
participants | 18

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the study, ie; from screening till the last day of the follow up period, an average of 14 weeks.
Arm/Group | 20% to 30% Salicylic Acid Peels + 4% Hydroquinone Cream
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20% to 30% Salicylic Acid Peels + 4% Hydroquinone Cream (N=20)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4)
Burning (Skin and subcutaneous tissue disorders) | 4 (4)
Peeling (Skin and subcutaneous tissue disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Two subjects did not complete the study were unable to come in for visits because of scheduling difficulties and had no adverse effects at the time of discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-10-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT00616239/Prot_SAP_000.pdf